CLINICAL TRIAL: NCT01851811
Title: To Examine the Correlation Between Continuous Positive Airway Pressure (CPAP) and the Timing of Last Meal Before Bed Time.
Brief Title: Correlation Between CPAP Compliance and Food Intake Timing
Acronym: TLMECC
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00000359
Record Dates: First submitted 2013-05-07; First posted 2013-05-13 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite widespread agreement that continuous positive airway pressure is effective therapy for obstructive sleep apnea, it is estimated that 50% of patients recommended for therapy are noncompliant 1 year later. Nasal continuous positive airway pressure (CPAP) is the most definitive medical therapy for obstructive sleep apnea (OSA). Many patients have difficulty tolerating nasal CPAP due to nasal airway problems, mouth leak, and general discomfort from the mask and headgear. Interventions to improve compliance in such patients have not been studied. The investigators plan to further evaluate the usage of CPAP and identify if the timing of last meal before bedtime affects the compliance and tolerance of CPAP.

DETAILED DESCRIPTION:
OSA is a chronic disorder characterized by frequent reduction and/or cessation of inspiratory airflow during sleep, with resulting hypoxemia and hypercapnia that are terminated by arousals. This pattern of repetitive arousals and nocturnal hypoxemia leads to disruption of sleep architecture and daytime hyper-somnolence as well as a multitude of neurobehavioral and cardiopulmonary derangements. All patients diagnosed with OSA should be instructed to undergo behavioral changes such as weight loss, avoidance of alcohol and sedatives, sleeping on the side and improvement in sleep hygiene, such as keeping a regular sleep schedule and getting an adequate amount of sleep. Continuous Positive Airways Pressure (CPAP) is currently considered to be the cornerstone of therapy for sleep apnea (OSA). However compliance with this treatment is frequently poor, which may lead to ongoing symptoms of sleep disruption, daytime sleepiness and poor waking cognitive function. Mechanical and psychological/educational interventions have been proposed to try to increase the hours of use of CPAP therapy. In older male patients with OSA, compliance with CPAP therapy is associated with attendance at a patient CPAP education and support group. Resolution of symptoms with therapy also appears to be associated with enhanced compliance. Some studies suggest that there is no direct causal relationship between OSA and gastro esophageal reflux disease (GERD). The investigators hypothesize that the compliance and tolerance to CPAP is affected with the timing of last meal before bedtime and this may also affect the symptoms of GERD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Obstructive Sleep Apnea.
* Patients on CPAP therapy
* Patients older than 21 years

Exclusion Criteria:

-Patients not on CPAP therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the HUMC who are diagnosed with sleep apnea will be determined through screening charts.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Correlation between Continuous Positive Airway Pressure (CPAP) and the timing of last meal before bed time | 12 months
  Questionnaires will be used to determine correlation

CONTACTS AND LOCATIONS:
Overall Officials: Susan Zafarlotfi, PhD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States